CLINICAL TRIAL: NCT05776498
Title: Clinical and Radiographic Evaluation of Immediate Implant Placement Using Dual Zone Approach Versus Connective Tissue Graft: A Randomized Clinical Trial
Brief Title: Evaluation of Immediate Implant Placement Using Dual Zone Approach Versus Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDCE.N3
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Immediate Dental Implants
Keywords: Immediate dental implants; anterior maxilla; esthetic zone; connective tissue graft; dual zone technique; bone graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement with particulate bone graft using the dual zone technique. (Experimental): immediate implant placement with particulate bone graft using the dual zone technique.
  Interventions: Procedure: immediate implant placement with particulate bone graft using the dual zone technique.
- immediate implant placement with connective tissue grafting (Experimental): immediate implant placement with connective tissue grafting
  Interventions: Procedure: immediate implant placement with connective tissue grafting

INTERVENTIONS:
Procedure: immediate implant placement with particulate bone graft using the dual zone technique. — Tooth extraction and immediate implant placement as mentioned, then particulate bone graft will be packed in the gap between the implant and the buccal plate of bone and the tissue (dual zone), then will be covered by a customized healing abutment.
  Arms: immediate implant placement with particulate bone graft using the dual zone technique.
Procedure: immediate implant placement with connective tissue grafting — Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supraperiosteal partial dissection pouch prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place. Followed by customized healing abutment.
  Arms: immediate implant placement with connective tissue grafting

SUMMARY:
Tooth extraction is followed by ridge alteration and soft tissue collapse and recession. Different strategies were proposed to limit this collapse however, the ability of these techniques to mimic the original soft tissue level and to maintain long term stability is unclear (Slagter et al., 2014). Using customized contoured healing abutments at the time of immediate implant placement is a treatment modality to improve esthetics by maintaining the soft tissue level and contour (Ruales-Carrera et al, 2019, Perez et al, 2020). Using connective tissue grafts has been suggested to enhance and maintain soft tissue stability, however, the effect of the combined procedures for maintenance of the soft tissue morphology compared to customized healing abutments alone remains unclear (Atieh et al, 2019). In patients with non-restorable teeth in the esthetic zone, will the use of bone grafts to the dual zone with customized healing abutment vs the use of connective tissue graft with customized healing abutment in immediately placed implants shows better buccal contour avoiding horizontal collapse?

ELIGIBILITY:
Inclusion criteria:

Patient-related criteria:

* Adults at or above the age of 18.
* Non-restorable maxillary anterior or premolar tooth requiring extraction and needed an implant placing therapy.
* The failing tooth will have adjacent and opposing natural teeth.
* Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration.
* Able to tolerate surgical periodontal procedures.
* Full mouth plaque and bleeding scores less than 20%.
* Compliance with the maintenance program.
* Provide informed consent.
* Accepts the one-year follow-up period.

Teeth related criteria:

* Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
* Intact socket wall before the extraction, buccal bone thickness ≤1mm assessed by CBCT.
* Sufficient apical bone to place an immediate implant with minimum primary stability of 30Ncm.

Exclusion criteria:

* Patients diagnosed with periodontal diseases.
* Current or previous smokers.
* Pregnant and lactating females.
* Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking IV Bis-phosphonates for treatment of osteoporosis.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with parafunctional habits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
pink esthetic score (PES) | 3 months after crown placement
  To evaluate the pink esthetic score 1-14 score

SECONDARY OUTCOMES:
Volumetric analysis of buccal contour | 6 months
  3D viewer soft tissue; mm changes in the buccal soft tissue contour in comparison to the original ones, at 2,4 and 6 mm from the pre-operative gingival margin
Mid-facial recession | 1 year
  3D viewer soft tissue
Interdental papilla | 1 year
  3D viewer soft tissue
Horizontal labio-palatal bone width | 1 year
  CBCT cone beam CT
Bone formed labial to the implant | 1 year
  CBCT cone beam CT
gingival biotype | 1 year
  thickness in millimeters mm

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Ghallab, PhD, Study Director — Professor of Oral Medicine & Periodontology
Locations (1):
- International Dental Continuing Education, Cairo, Egypt